CLINICAL TRIAL: NCT01091870
Title: Sildenafil for Prevention of Cerebral Vasospasm Secondary to Subarachnoid Haemorrhage - Phase II Randomized Clinical Trial
Brief Title: Sildenafil for Prevention of Cerebral Vasospasm
Acronym: SIPCEVA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Absence of inclusion criteria
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIPCEVA; 09453 (Other: Etics Comitee of Hospital de Clínicas de Porto Alegre)
Record Dates: First submitted 2010-03-17; First posted 2010-03-24 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm; Rupture of Intracranial Aneurysm
Keywords: Aneurysm; Vasospasm; sildenafil; Viagra
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Aneurysm | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo: soluble blue pigment (Placebo Comparator): Soluble blue pigment for placebo controlling.
  Interventions: Drug: Placebo
- Sildenafil, 75mg daily (Experimental): Sildenafil citrate, 75 mg daily divided in 3 doses. From third to 14th day after subarachnoid hemorrhage.
  Interventions: Drug: Sildenafil Citrate, 25 mg, 3 times a day.
- Sildenafil, 150 mg daily (Experimental): Sildenafil citrate, 150 mg daily divided in 3 doses from third to 14th day after subarachnoid hemorrhage.
  Interventions: Drug: Sildenafil Citrate 50 mg, 3 times a day

INTERVENTIONS:
Drug: Placebo — Soluble blue pigment, 3 times a day, from the third to the 14th day after subarachnoid hemorrhage.
  Arms: Placebo: soluble blue pigment
Drug: Sildenafil Citrate, 25 mg, 3 times a day. — Sildenafil Citrate 25 mg, 3 times a day (TID)from the third to the 14 day after subarachnoid hemorrhage.
  Other Names: Viagra
  Arms: Sildenafil, 75mg daily
Drug: Sildenafil Citrate 50 mg, 3 times a day — Sildenafil Citrate 25 mg, 3 times a day (TID)from the third to the 14 day after subarachnoid hemorrhage.
  Other Names: Viagra
  Arms: Sildenafil, 150 mg daily

SUMMARY:
A Randomized Clinical Trial with security and dose testing of Sildenafil Citrate in patients with subarachnoid hemorrhage due to a rupture of a cerebral aneurism for prevention of cerebral vasospasm. The cerebral vasospasm is a decrease in blood flow that occurs when the intracranial vessels lose their capability of self-control of dilations and contractions. Patients with subarachnoid hemorrhage without neurological deficits who underwent endovascular or surgical correction of the aneurysm can participate in this trial. They will be randomized to a daily doses of 75 mg of Sildenafil, 150 mg of Sildenafil or Placebo from the third to the 14th day post bleeding. Today there is no proven clinical treatment for prevention of cerebral vasospasm.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 20 and 80 years old
* Subarachnoid hemorrhage confirmed by CT with Fisher III or IV criteria (blood in cisterns larger than 1 mm with or without blood in the ventricular system).
* Aneurysm detected in the conventional angiography, or angio-CT or angio - MRI.
* Patient underwent surgery for clipping or endovascular treatment in the first 72 hours after the ictus.
* Consent form signed by the patient or legal responsible.

Exclusion Criteria:

* Patient (or legal responsible) refuses to participate.
* Impossibility to collect consent form.
* Hemodynamical instability.
* Previous cardiac ischemic disease.
* History of cardiac arrhythmia within the last 6 months.
* History of Retinitis Pigmentosa.
* Previous use of drugs witch can interact with sildenafil (specially nitrates).
* Pregnancy.
* Known hypersensibility to Sildenafil.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
New neurological Deficit | From third to 14th day post subarachnoid hemorrhage
  Development of clinical symptoms suggestive of vasospasm, which are: afasia, hemiparesis, disorientation, or worsening of consciousness without hydrocephalus or expanding cloth. To access level of consciousness we will use the Glasgow Coma Scale.

SECONDARY OUTCOMES:
Transcranial Ecodoppler | From the third to the 14th day after subarachnoid hemorrhage
  Signs of vasospasm in in transcranial ecodoppler.
Mortality | From the third to the 14th day before subarachnoid hemorrhage.
  General mortality (for any causes).
Side effects | From the third to the 14th day after subarachnoid hemorrhage.
  Drug side effect: hypotension, visual blurring, nasal congestion, angina pectoris, asthma crisis, AV block, digestive bleeding, and priapism.
Time to discharge | From the third day after subarachnoid hemorrhage to discharge.
  Time to discharge (period of hospital stay).
Rankin Scale | At discharge from the hospital.
  Modified Rankin scale at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: André Cerutti Franciscatto, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre; Marco Antônio Stefani, DR, Study Director — Hospital de Clínicas de Porto Alegre; Ápio Martins Antunes, DR, Study Chair — Hospital de Clínicas de Porto Alegre; Thiago Torres de Ávila, MD, Study Chair — Hospital de Clínicas de Porto Alegre; Mateus Lasta Beck, MD, Study Chair — Hospital de Clínicas de Porto Alegre; Mateus Franzói, MD, Study Chair — Hospital de Clínicas de Porto Alegre; Atahualpa Caue Strapasson, MD, Study Chair — Hospital de Clínicas de Porto Alegre; Sílvia Brustolin, DR, Study Chair — Hospital de Clínicas de Porto Alegre; Fabiane Backes, MD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Official Site of Hospital de Clínicas de Porto Alegre — http://www.hcpa.ufrgs.br